CLINICAL TRIAL: NCT04715490
Title: Effects of a Multimedia Symptom Management Program on Coping Strategies, Symptom Distress, Depressive Status, and Quality of Life in Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: Effects of a Multimedia Symptom Management Program on Quality of Life in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Fung-Wei Chang, Director, Head of Obstetrics and Gynecology, Clinical Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tri_20200114
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: multimedia; coping strategy; symptom distress; quality of life
MeSH Terms: conditions — Heart Failure | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Multimedia Symptom Management Program Intervention (Experimental): The program is composed of two parts: 1) a face-to-face presentation about the contents of the program, and 2) structured telephone support.
  Interventions: Other: The Multimedia Symptom Management Program Intervention
- Control group (Active Comparator): Participants in the control group will be provided with the HF handbook at the beginning of the 3-month period, and also will be received usual care, which included medical consultations, and two telephone calls.
  Interventions: Other: Control group

INTERVENTIONS:
Other: The Multimedia Symptom Management Program Intervention — The program is composed of two parts: 1) a face-to-face presentation about the contents of the program, and 2) structured telephone support. The first part of the program will be conducted in the cardiology outpatient department. Participants will be instructed to read a HF handbook.
  The second part of the program, structured telephone support, allowed the nurses to maintain contact with the participants in order to follow their progress. The participants will be scheduled to receive eight telephone coaching calls over a 3-month period.
  Arms: The Multimedia Symptom Management Program Intervention
Other: Control group — The control group will be provided with the HF handbook at the beginning of the 3-month period, and also will be received usual care, which included medical consultations, and two telephone calls.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a Multimedia Symptom Management Program on increasing coping strategies, reducing symptom distress and depression, and improving HRQoL in patients with HF.

DETAILED DESCRIPTION:
Design A single-blind two-group longitudinal experimental study will be conducted to compare a Multimedia Symptom Management Program with a usual care.

After receiving informed consents, participants will be randomly assigned to intervention and control groups at a 1:1 ratio. The intervention group will receive a Multimedia Symptom Management Program; the control group will receive usual care. Outcomes from four self-report questionnaires at 1 month and 3 months after initiating the intervention will be compared to baseline assessments. Outcome measurements include the following parameters: 28-item Brief COPE, Cardiac Symptom Survey (CSS), Beck Depression Inventory-II (BDI-II), and Minnesota Living with Heart Failure Questionnaire (MLHFQ).

Inclusion and exclusion criteria The inclusion criteria are: (1) those who are ≥20 years old and HF diagnosed by a cardiology specialist, (2) have clear consciousness, (3) are fluent in Mandarin/Taiwanese. The exclusion criteria are: (1) diagnosed with any psychiatric disorder, (2) are addicting to drugs or alcohol at the time of the study, (3) are undergoing other psychotherapy during the study and (4) are refusing to participate in the study.

Recruitment Participants will be recruited from a cardiology outpatient clinic of a medical center in northern Taiwan. The study design and protocols had been reviewed and approved by the institutional review board of the participating hospital. At the content session, all assessments and procedures will be fully explained.

Assessment of eligibility and randomisation Participants will be considered eligible if they meet the inclusion criteria. All participants will be informed that they are able to withdraw from the study at any time. Before randomisation, participants will be asked to answer five questionnaires. The questionnaires include demographic characteristics, 28-item Brief COPE, Cardiac Symptom Survey (CSS), Beck Depression Inventory-II (BDI-II), and Minnesota Living with Heart Failure Questionnaire (MLHFQ). Participants will be randomly assigned to either the intervention group or the control group at a 1:1 ratio; randomization will be performed with the use of a computer-generated randomization scheme (SPSS software Version 23.0).

Blinding Participants will be randomly assigned to either the Multimedia Symptom Management Program or medical consultation and usual care. Random assignment will be performed by a person who are not involved in the study. The outcome evaluator will be blinded to the assigned condition of the participants.

Intervention Participants will be randomly assigned to the Multimedia Symptom Management Program Intervention group or the control group using SPSS software (Version 23.0).

The Multimedia Symptom Management Program Intervention The program is composed of two parts: 1) a face-to-face presentation about the contents of the program, and 2) structured telephone support. The first part of the program will be conducted in the cardiology outpatient department. Participants will be instructed to read a HF handbook. In addition, they will also be provided with multimedia symptom management instruction through a live-action feature film on a DVD, which will be designed and produced by the researchers to help familiarize patients with the symptoms and characteristics of HF, how to perform self-evaluations, and ways to manage symptoms of HF. After the conclusion of the face-to-face presentation, we will ensure that participants have fully comprehended all instructions with the return demonstration method, in which participants had reviewed the HF handbook and multimedia symptom management DVD at home and will be encouraged to review management of their symptoms daily.

The second part of the program, structured telephone support, allowed the nurses to maintain contact with the participants in order to follow their progress. The participants will be scheduled to receive eight telephone coaching calls over a 3-month period. In the first month, participants will receive telephone coaching calls every week. Through the phone calls, the nurse clinician will try to sustain the participants' symptom management knowledge and skills by encouraging them to discuss what they had learned from the DVD to discuss how they had managed their symptoms. Subsequent telephone counselling calls will be conducted every 2 weeks in the second and third months to follow their situations and assist them in dealing with any health problems.

Control group Participants in the control group will be provided with the HF handbook at the beginning of the 3-month period, and also will be received usual care, which included medical consultations, and two telephone calls.

Outcomes measurements Primary outcome Health-related quality of life (HRQoL): The 21-item Minnesota Living with Heart Failure Questionnaire (MLHFQ) is used to measure HRQoL in adult patients with HF. A 6-point Likert scale is used to score the impact on HRQoL from 0 = "No effect" to 5 = "Severe effect". Total scores range from 0 to 105, with higher scores indicating a worse HRQoL. The Cronbach's alpha coefficient of MLHFQ was 0.92.

Secondary outcome Brief COPE: The 28-item Brief COPE self-report questionnaire measure strategies participants use for coping. The Brief-COPE is divided into approach coping, in which individuals actively seek resources to deal with their health problems; and avoidance coping, in which individuals attempt to divert attention away from events. Higher scores indicate greater use of the specific coping strategy.

Cardiac Symptom Survey (CSS): CSS is originally used as a tool to assess symptoms of patients undergoing coronary artery bypass surgery, assessed symptom distress. In this study, we only assessed only the 20 items for frequency and severity of symptoms. We obtained permission from Dr. L. J. Nieveen to change the wording of one item, "surgery pain", to "activity intolerance".

Beck Depression Inventory-II (BDI-II): BDI-II is used to measure the depressive status of participants. The self-report questionnaire asks about symptoms of depression over a 2-week period. Higher total scores indicating a more severe of depressive status: 0-13 = normal; 14-29 = mild; 28-28 = moderate; and 29-63 = severe depressive status.

Statistical analysis We will use descriptive statistics (mean, standard deviation, frequency and percentage) to analyse participant characteristics and primary outcomes. The initial differences between groups for demographic characteristics, symptom distress, coping strategies, depressive status, and HRQoL will be examined with independent t-tests and Chi-square analysis. Effects of the Multimedia Symptom Management Program on symptom distress, coping strategies, depressive status and HRQoL in patients with HF will be analysed using generalized estimating equations (GEE). The significance will be defined as a two-tailed P-value of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. those who are ≥20 years old and HF diagnosed by a cardiology specialist
2. have clear consciousness
3. are fluent in Mandarin/Taiwanese.

Exclusion Criteria:

1. diagnosed with any psychiatric disorder
2. are addicting to drugs or alcohol at the time of the study
3. are undergoing other clinical trial during the study
4. are refusing to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | Change from quality of life at 3 months

SECONDARY OUTCOMES:
28-item Brief COPE | Change from coping strategy at 3 months
Cardiac Symptom Survey Questionnaire | Change from symptom distress at 3 months
Beck Depression Inventory-II | Change from depressive status at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Kao, PHD, Study Director — Taiwan Nurses Association

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li CC, Shun SC. Understanding self care coping styles in patients with chronic heart failure: A systematic review. Eur J Cardiovasc Nurs. 2016 Feb;15(1):12-9. doi: 10.1177/1474515115572046. Epub 2015 Feb 13. PMID 25681369
- [Result] Gellis ZD, Kenaley BL, Ten Have T. Integrated telehealth care for chronic illness and depression in geriatric home care patients: the Integrated Telehealth Education and Activation of Mood (I-TEAM) study. J Am Geriatr Soc. 2014 May;62(5):889-95. doi: 10.1111/jgs.12776. Epub 2014 Mar 21. PMID 24655228
- [Result] Feltner C, Jones CD, Cene CW, Zheng ZJ, Sueta CA, Coker-Schwimmer EJ, Arvanitis M, Lohr KN, Middleton JC, Jonas DE. Transitional care interventions to prevent readmissions for persons with heart failure: a systematic review and meta-analysis. Ann Intern Med. 2014 Jun 3;160(11):774-84. doi: 10.7326/M14-0083. PMID 24862840
- [Result] Abbasi A, Najafi Ghezeljeh T, Ashghali Farahani M, Naderi N. Effects of the self-management education program using the multi-method approach and multimedia on the quality of life of patients with chronic heart failure: A non-randomized controlled clinical trial. Contemp Nurse. 2018 Aug-Oct;54(4-5):409-420. doi: 10.1080/10376178.2018.1538705. Epub 2018 Oct 31. PMID 30381006
- [Result] Li CC, Chang SR, Shun SC. The self-care coping process in patients with chronic heart failure: A qualitative study. J Clin Nurs. 2019 Feb;28(3-4):509-519. doi: 10.1111/jocn.14640. Epub 2018 Aug 28. PMID 30091501
- [Result] Malik AH, Malik SS, Aronow WS; MAGIC (Meta-analysis And oriGinal Investigation in Cardiology) investigators. Effect of home-based follow-up intervention on readmissions and mortality in heart failure patients: a meta-analysis. Future Cardiol. 2019 Sep;15(5):377-386. doi: 10.2217/fca-2018-0061. Epub 2019 Sep 10. PMID 31502879
- [Result] Nes LS, Segerstrom SC. Dispositional optimism and coping: a meta-analytic review. Pers Soc Psychol Rev. 2006;10(3):235-51. doi: 10.1207/s15327957pspr1003_3. PMID 16859439
- [Result] Piamjariyakul U, Thompson NC, Russell C, Smith CE. The effect of nurse-led group discussions by race on depressive symptoms in patients with heart failure. Heart Lung. 2018 May-Jun;47(3):211-215. doi: 10.1016/j.hrtlng.2018.02.005. Epub 2018 Mar 30. PMID 29606370
- [Result] Mizukawa M, Moriyama M, Yamamoto H, Rahman MM, Naka M, Kitagawa T, Kobayashi S, Oda N, Yasunobu Y, Tomiyama M, Morishima N, Matsuda K, Kihara Y. Nurse-Led Collaborative Management Using Telemonitoring Improves Quality of Life and Prevention of Rehospitalization in Patients with Heart Failure. Int Heart J. 2019 Nov 30;60(6):1293-1302. doi: 10.1536/ihj.19-313. Epub 2019 Nov 15. PMID 31735786
- [Result] Smith CE, Piamjariyakul U, Dalton KM, Russell C, Wick J, Ellerbeck EF. Nurse-Led Multidisciplinary Heart Failure Group Clinic Appointments: Methods, Materials, and Outcomes Used in the Clinical Trial. J Cardiovasc Nurs. 2015 Jul-Aug;30(4 Suppl 1):S25-34. doi: 10.1097/JCN.0000000000000255. PMID 25774836
- [Result] Oyanguren J, Latorre Garcia PM, Torcal Laguna J, Lekuona Goya I, Rubio Martin S, Maull Lafuente E, Grandes G. Effectiveness and Factors Determining the Success of Management Programs for Patients With Heart Failure: A Systematic Review and Meta-analysis. Rev Esp Cardiol (Engl Ed). 2016 Oct;69(10):900-914. doi: 10.1016/j.rec.2016.05.012. English, Spanish. PMID 27692124
- [Result] Mayer RE. Applying the science of learning to medical education. Med Educ. 2010 Jun;44(6):543-9. doi: 10.1111/j.1365-2923.2010.03624.x. PMID 20604850
- [Result] Tomavo S, Dubremetz JF, Entzeroth R. Characterization of a surface antigen of Eimeria nieschulzi (Apicomplexa, Eimeriidae) sporozoites. Parasitol Res. 1989;75(5):343-7. doi: 10.1007/BF00931128. PMID 2657714
- [Result] Gagne M, Legault C, Boulet LP, Charbonneau L, Lemyre M, Giguere AMC, Poirier P. Impact of adding a video to patient education on quality of life among adults with atrial fibrillation: a randomized controlled trial. Patient Educ Couns. 2019 Aug;102(8):1490-1498. doi: 10.1016/j.pec.2019.03.015. Epub 2019 Mar 31. PMID 30956021
- [Result] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Result] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Result] Franks HM, Roesch SC. Appraisals and coping in people living with cancer: a meta-analysis. Psychooncology. 2006 Dec;15(12):1027-37. doi: 10.1002/pon.1043. PMID 16602072
- [Result] Nieveen JL, Zimmerman LM, Barnason SA, Yates BC. Development and content validity testing of the Cardiac Symptom Survey in patients after coronary artery bypass grafting. Heart Lung. 2008 Jan-Feb;37(1):17-27. doi: 10.1016/j.hrtlng.2006.12.002. PMID 18206523